CLINICAL TRIAL: NCT02848339
Title: Aspirin DesensitizAtion in PatienTs With Coronary artEry Disease: Results of a Multi Center Registry: the ADAPTED Registry
Brief Title: Aspirin Desensitization Registry in Patients With Aspirin Hypersensitivity
Acronym: ADAPTED
Status: Completed | Type: Observational
Sponsor: Italian Society of Cardiology (Other)
Responsible Party: Principal Investigator, Roberta Rossini, MD Ph D, Italian Society of Cardiology
Other Study IDs: GISE
Record Dates: First submitted 2016-07-22; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Aspirin Hypersensitivity
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: aspirin — aspirin desensitization

SUMMARY:
Data about aspirin desensitization for patients with coronary artery disease undergoing percutaneous coronary intervention are sparse.

This is a prospective, multicenter, observational study including 7 italian centers, to assess safety and feasibility of a standard desensitization protocol in patients with aspirin sensitivity undergoing coronary angiography. Patients with history of aspirin sensitivity undergoing coronary angiography are prospectively enrolled.All patients underwent the desensitization procedure with six sequential doses of aspirin (1, 5, 10, 20, 40, and 100 mg) administered orally at predefined intervals, with the procedure lasting 5.5 hours.All patients are followed for desensitization procedure success, description of reactions due to the desensitization procedure, and in hospital major adverse cardiac events (MACE). All patients are also followed-up for 12 months in order to assess their long-term risk of MACE, compliance with ASA therapy, and late occurrence of side reactions due to ASA sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* history of aspirin hypersensitivity
* acute coronary syndrome or known/suspected stable coronary artery disease
* intent to undergo percutaneous coronary intervention

Exclusion Criteria:

* withdrawal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of aspirin hypersensitivity presenting with either an acute coronary syndrome or known/suspected stable coronary artery disease scheduled for coronary angiography with intent to undergo PCI
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2010-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with successful desensitization procedure | 12 months
  All patients are followed for desensitization procedure success, description of reactions due to the desensitization procedure.
Major adverse cardiac events | 12 months
  Percentage of patients with an adverse cardiac event (cardiac death, myocardial infarction, stent thrombosis, stroke, destabilizing symptoms leading to hospitalization

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Rossini R, Iorio A, Pozzi R, Bianco M, Musumeci G, Leonardi S, Lettieri C, Bossi I, Colombo P, Rigattieri S, Dossena C, Anzuini A, Capodanno D, Senni M, Angiolillo DJ. Aspirin Desensitization in Patients With Coronary Artery Disease: Results of the Multicenter ADAPTED Registry (Aspirin Desensitization in Patients With Coronary Artery Disease). Circ Cardiovasc Interv. 2017 Feb;10(2):e004368. doi: 10.1161/CIRCINTERVENTIONS.116.004368. PMID 28193678